CLINICAL TRIAL: NCT07075302
Title: Comparison of Postoperative Morphine Requirements Between an Opioid-Based and an Opioid-Free Anesthesia Technique in Morbidly Obese Patients Undergoing Bariatric Surgery
Brief Title: OFA vs OBA in Bariatric Surgery
Acronym: OFA VS OBA1
Status: Completed | Type: Observational
Sponsor: Hospital HM Nou Delfos (Other)
Responsible Party: Principal Investigator, HIPÓLITO LABANDEYRA GONZALEZ, Anesthesiologist, Hospital HM Nou Delfos
Other Study IDs: 25.04.2517-GHM
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Postoperative Pain; Bariatric Surgery; Opioid-free Anesthesia
Keywords: Opioid-Free Anesthesia; Bariatric Surgery; opioid-based anesthesia; morphine consumption; TIVA; multimodal analgesia
MeSH Terms: conditions — Obesity; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OFA Group: Patients who received opioid-free total intravenous anesthesia (TIVA) for bariatric surgery, including propofol, lidocaine, ketamine, dexmedetomidine and magnesium, with no intraoperative opioids.
- OBA Group: Patients who received opioid-based total intravenous anesthesia (TIVA) for bariatric surgery, including propofol and intraoperative opioids such as fentanyl, remifentanil and morphine, following standard practice.

SUMMARY:
This study compares two different anesthesia techniques in patients with obesity undergoing bariatric surgery: one that includes opioids (OBA), and one that avoids them completely (OFA). The main goal is to determine whether avoiding opioids during surgery leads to lower postoperative morphine requirements and fewer side effects. Researchers reviewed medical records of 70 patients who had bariatric surgery between June 2022 and December 2023 at a hospital in Spain. The study evaluates pain levels, sedation, complications, and total morphine use in the first 48 hours after surgery.

DETAILED DESCRIPTION:
This is a single-center, retrospective, observational cohort study conducted at Hospital HM Nou Delfos (Barcelona, Spain). The aim is to compare postoperative opioid requirements and outcomes in patients with morbid obesity undergoing laparoscopic bariatric surgery, according to the intraoperative anesthesia technique used.

Two anesthetic strategies were evaluated:

Opioid-Free Anesthesia (OFA): Total intravenous anesthesia (TIVA) without opioids, using agents such as propofol, ketamine, dexmedetomidine, lidocaine and magnesium.

Opioid-Based Anesthesia (OBA): TIVA including opioids, following institutional standards.

Medical records of 70 patients (35 in each group) who underwent surgery between June 2022 and December 2023 were analyzed. Key data extracted included demographics, surgical duration, anesthetic drugs used, intraoperative complications, pain scores (VAS at 1, 2, 4, 24, and 48 hours), sedation levels (RAMSAY scale), adverse effects (e.g., nausea, vomiting, ileus, hypotension), and morphine consumption.

The primary outcome is total morphine use within the first 48 hours postoperatively. Secondary outcomes include pain scores, adverse events, time to awakening, and hospital length of stay. Statistical analysis was performed using descriptive and inferential methods, including regression models adjusted for age, sex, BMI, and comorbidities.

This study provides real-world evidence on the clinical impact of opioid-free anesthesia in bariatric patients, aiming to improve perioperative safety and enhance postoperative recovery.

ELIGIBILITY:
Inclusion Criteria Age between 18 and 65 years

Body Mass Index (BMI) ≥ 30 kg/m²

ASA physical status II or III

Underwent laparoscopic bariatric surgery under general anesthesia at HM Nou Delfos

Surgery performed between June 1, 2022 and December 31, 2023

Exclusion Criteria Pregnancy or breastfeeding

Chronic pain patients on high-dose opioids

Known allergy to any anesthetic drug used in the study

Severe hepatic (e.g., cirrhosis with portal hypertension) or renal insufficiency

Untreated coagulopathy

Active alcohol or drug abuse

Uncontrolled or severe psychiatric illness

Intraoperative complications requiring deviation from planned anesthetic technique

Postoperative morphine use exceeding institutional norms for bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-65 years) with obesity (BMI ≥ 30 kg/m²) classified as ASA II-III, who underwent laparoscopic bariatric surgery under general anesthesia at HM Nou Delfos between June 2022 and December 2023. Patients were retrospectively assigned to one of two groups based on the anesthetic technique used: opioid-free anesthesia (OFA) or opioid-based anesthesia (OBA).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Total postoperative morphine consumption (mg) | From 0 to 48 hours after surgery
  Cumulative amount of morphine (in milligrams) administered within the first 48 hours after surgery, as recorded in the post-anesthesia care unit and inpatient medical records.

SECONDARY OUTCOMES:
Pain intensity (VAS) | At 1, 2, 4, 24, and 48 hours postoperatively
  Pain evaluated using the Visual Analog Scale (VAS) from 0 (no pain) to 10 (worst imaginable pain), both at rest and with movement.
Sedation level (RAMSAY scale) | From 0 to 48 hours after surgery
  Sedation assessed using the Ramsay Sedation Scale, ranging from 1 (anxious/agitated) to 6 (no response to stimuli).
Incidence of adverse events | Up to 48 hours after surgery
  Number of patients experiencing side effects such as nausea, vomiting, pruritus, hypotension, bradycardia, ileus, or urinary retention.
Length of hospital stay | From surgery until discharge (up to 7 days)
  Total duration of hospital stay in days, calculated from the day of surgery to discharge date.
Time to awakening | Intraoperative period until recovery (measured at end of surgery)
  Time in minutes from the end of surgery until patient opens eyes or responds to verbal commands.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Contreras-Pérez, Anesthesiologist, Principal Investigator — Hospital HM NouDelfos
Locations (1):
- Hospital HM Nou Delfos, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
This is a retrospective study involving patient health records. Due to ethical and privacy regulations, individual participant data cannot be shared publicly. Access is restricted to the research team as approved by the ethics committee.

REFERENCES:
- [Background] Kumar A, Kohli A. Comeback of ketamine: resurfacing facts and dispelling myths. Korean J Anesthesiol. 2021 Apr;74(2):103-114. doi: 10.4097/kja.20663. Epub 2021 Jan 11. PMID 33423410
- [Background] Brannian JD, McCulloh DH. Gonadotropin control of follicle and oocyte maturation: implications for ovulation induction. S D J Med. 1995 Oct;48(10):335-9. PMID 7502015
- [Background] Roesslein M, Chung F. Obstructive sleep apnoea in adults: peri-operative considerations: A narrative review. Eur J Anaesthesiol. 2018 Apr;35(4):245-255. doi: 10.1097/EJA.0000000000000765. PMID 29300271
- [Background] Hofer RE, Sprung J, Sarr MG, Wedel DJ. Anesthesia for a patient with morbid obesity using dexmedetomidine without narcotics. Can J Anaesth. 2005 Feb;52(2):176-80. doi: 10.1007/BF03027725. PMID 15684259
- [Background] Mantz J, Josserand J, Hamada S. Dexmedetomidine: new insights. Eur J Anaesthesiol. 2011 Jan;28(1):3-6. doi: 10.1097/EJA.0b013e32833e266d. PMID 20881501
- [Background] Candiotti KA, Bergese SD, Bokesch PM, Feldman MA, Wisemandle W, Bekker AY; MAC Study Group. Monitored anesthesia care with dexmedetomidine: a prospective, randomized, double-blind, multicenter trial. Anesth Analg. 2010 Jan 1;110(1):47-56. doi: 10.1213/ane.0b013e3181ae0856. Epub 2009 Aug 27. PMID 19713256
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Fuchs-Buder T, Schmartz D, Baumann C, Hilt L, Nomine-Criqui C, Meistelman C, Brunaud L. Deep neuromuscular blockade improves surgical conditions during gastric bypass surgery for morbid obesity: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jul;36(7):486-493. doi: 10.1097/EJA.0000000000000996. PMID 30985536
- [Background] Ingrande J, Lemmens HJ. Dose adjustment of anaesthetics in the morbidly obese. Br J Anaesth. 2010 Dec;105 Suppl 1:i16-23. doi: 10.1093/bja/aeq312. PMID 21148651
- [Background] Raveendran R, Wong J, Singh M, Wong DT, Chung F. Obesity hypoventilation syndrome, sleep apnea, overlap syndrome: perioperative management to prevent complications. Curr Opin Anaesthesiol. 2017 Feb;30(1):146-155. doi: 10.1097/ACO.0000000000000421. PMID 27792079
- [Background] Schumann R, Shikora SA, Sigl JC, Kelley SD. Association of metabolic syndrome and surgical factors with pulmonary adverse events, and longitudinal mortality in bariatric surgery. Br J Anaesth. 2015 Jan;114(1):83-90. doi: 10.1093/bja/aeu362. Epub 2014 Oct 13. PMID 25311316
- [Background] Sultana A, Torres D, Schumann R. Special indications for Opioid Free Anaesthesia and Analgesia, patient and procedure related: Including obesity, sleep apnoea, chronic obstructive pulmonary disease, complex regional pain syndromes, opioid addiction and cancer surgery. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):547-560. doi: 10.1016/j.bpa.2017.11.002. Epub 2017 Nov 16. PMID 29739543
- [Background] de Raaff CAL, de Vries N, van Wagensveld BA. Obstructive sleep apnea and bariatric surgical guidelines: summary and update. Curr Opin Anaesthesiol. 2018 Feb;31(1):104-109. doi: 10.1097/ACO.0000000000000542. PMID 29176373
- [Background] Malo-Manso A, Ramirez-Aliaga M, Sepulveda-Haro E, Diaz-Crespo J, Escalona-Belmonte JJ, Guerrero-Orriach JL. Opioid-free anesthesia for open radical cystectomy in morbid obesity. Rev Esp Anestesiol Reanim (Engl Ed). 2021 Sep 23:S0034-9356(21)00134-1. doi: 10.1016/j.redar.2021.03.007. Online ahead of print. English, Spanish. PMID 34565571
- [Background] Al-Hasani R, Bruchas MR. Molecular mechanisms of opioid receptor-dependent signaling and behavior. Anesthesiology. 2011 Dec;115(6):1363-81. doi: 10.1097/ALN.0b013e318238bba6. PMID 22020140
- [Background] Kanjhan R. Opioids and pain. Clin Exp Pharmacol Physiol. 1995 Jun-Jul;22(6-7):397-403. doi: 10.1111/j.1440-1681.1995.tb02029.x. PMID 8582088
- [Background] Weiner SG, Malek SK, Price CN. The Opioid Crisis and Its Consequences. Transplantation. 2017 Apr;101(4):678-681. doi: 10.1097/TP.0000000000001671. No abstract available. PMID 28323774
- [Background] Burke DS. Forecasting the opioid epidemic. Science. 2016 Nov 4;354(6312):529. doi: 10.1126/science.aal2943. No abstract available. PMID 27811241
- [Background] Frauenknecht J, Kirkham KR, Jacot-Guillarmod A, Albrecht E. Analgesic impact of intra-operative opioids vs. opioid-free anaesthesia: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):651-662. doi: 10.1111/anae.14582. Epub 2019 Feb 25. PMID 30802933
- [Background] Chlif M, Keochkerian D, Choquet D, Vaidie A, Ahmaidi S. Effects of obesity on breathing pattern, ventilatory neural drive and mechanics. Respir Physiol Neurobiol. 2009 Sep 30;168(3):198-202. doi: 10.1016/j.resp.2009.06.012. Epub 2009 Jun 24. PMID 19559105